CLINICAL TRIAL: NCT03104751
Title: Neurodevelopment in Infants With Complex Congenital Heart Defects
Status: Completed | Type: Observational
Sponsor: Ohio State University (Other)
Collaborators: American Heart Association (Other); Nationwide Children's Hospital (Other)
Responsible Party: Principal Investigator, Jill Heathcock, Associate Professor, Ohio State University
Other Study IDs: 2015N0040
Record Dates: First submitted 2017-03-27; First posted 2017-04-07 (Actual); Last update posted 2021-02-24 (Actual); Status verified 2021-02

CONDITIONS: Complex Congenital Heart Defect
Keywords: Complex Congenital Heart Defect; Infants

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Infants with Complex Congenital Heart Defect: Infants diagnosed a Complex Congenital Heart Defect
- Comparison/Healthy Infants: Infants born without genetic syndromes or cardiac condition.

SUMMARY:
The primary goal of this study is to systematically describe early neurodevelopment using a complementary set of observational and neurophysiological measures that may predict cognitive and motor delays earlier than currently possible for infants with Complex Congenital Heart Disease (CCHD).

DETAILED DESCRIPTION:
The investigators' long-term goals are to develop a method of identifying infants likely to have adverse neurodevelopmental outcomes following neonatal treatment for CCHD and to develop and test interventions that can be applied early in infancy. The necessary first step is to systematically describe early neurodevelopment using a complementary set of observational and neurophysiological measures that may predict cognitive and motor delays earlier than currently possible for infants with CCHD. Each measure provides unique information about development and will include (1) neuroimaging for brain maturity and brain injury, (2) hair and fingernails for cortisol and saliva for immune system function, (3) heart rate variability (HRV) for autonomic nervous system function (ANS), (4) Bayley Scales of Infant Development (BSID-III) for cognitive and motor function, (5) a naturalistic play session incorporating kicking, general movement analysis, or the Test of Infant Motor Performance (TIMP) for motor development, and (6) the mobile paradigm for learning, memory, and task-specific coordination. The investigators will look at types of relationships among these measures within each time point for description of development and across each time point for prediction of development. The investigators' core hypotheses are that infants with CCHD will have measurable deficits in cognitive and motor development birth to ~ 6 months of age when compared with a healthy control group and that a typology developed from neurodevelopmental measures will reliably predict cognitive and motor delay in the first six months of life in infants with CCHD.

ELIGIBILITY:
Inclusion Criteria:

* at least 36 weeks gestational age
* diagnosed with a Complex Congenital Heart Defect
* have at least one English-speaking adult family member

Exclusion Criteria:

* presence of co-existing, non-cardiac congenital anomalies
* ongoing post-operative cardiac pacing

Ages: 1 Day to 30 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Participants are infants born with a complex congenital heart defect.Cardiac defects include, but are not be limited to: atrioventricular canal defect, double outlet right ventricle, hypoplastic left heart syndrome, interrupted aortic arch, pulmonary atresia, tetralogy of Fallot, and transposition of the great arteries.All participants are recruited from Nationwide Children's Hospital in Columbus, OH. Healthy infants will also be enrolled as a comparison group.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2016-06-30 (Actual); Primary Completion 2018-10-24 (Actual); Study Completion 2018-10-24 (Actual)

PRIMARY OUTCOMES:
Change in MRI (Magnetic Resonance Imaging) of brain - infants with CCHD only | 1 to 5 days days prior to surgery, 4-10 days after surgery, 6 months of age
  Brain MRI
Change in Test of Infant Motor Performance (TIMP) | 0-30 days, 3 months
  test of early motor development
Change in Mobile Paradigm | 3 months and 6 months
  Measure of learning, memory, and task-specific kicking coordination in infants
Change in Heart Rate Variability | 30 days, 3 months, 6 months
  Measure of autonomic nervous system function and development

SECONDARY OUTCOMES:
Bayley Scales of Motor Development | 3 months, 6 months
  The Bayley Scales of Infant and Toddler Development is an individually administered test designed to assess developmental functioning of infants and toddlers. The Bayley-III assesses development in five areas: cognitive, language, motor, social-emotional, and adaptive behavior.
Edinburgh Postnatal Depression Scale | 0-30 days, 3 months, 6 months
  self report survey to assess maternal depression
Infant-Toddler Quality of Life Questionnaire | 0-30 days, 3 months, 6 months
  self report survey to assess infant health status and physical and psychosocial functioning
State-Trait Anxiety Inventory | 0-30 days, 3 months, 6 months
  sefl report survey measure of anxiety

OTHER OUTCOMES:
Salivary cortisol | 0-30 days, 3 months, 6 months
  Saliva sample to measure snapshot of cortisol release
Hair cortisol | 0-30 days, 3 months, 6 months
  Hair cortisol provides a validated measure of intensity and course of stress exposure over time and is considered a proxy measure of total HPA activation
Fingernail cortisol | 0-30 days, 3 months, 6 months
  Fingernail sample to measure cortisol levels

CONTACTS AND LOCATIONS:
Overall Officials: Jill Heathcock, MPT, PhD, Principal Investigator — Ohio State University
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States

REFERENCES:
- [Derived] Tripathi T, Harrison TM, Simsic JM, Cabral TI, Heathcock JC. Screening and Evaluation of Neurodevelopmental Impairments in Infants Under 6 Months of Age with Congenital Heart Disease. Pediatr Cardiol. 2022 Mar;43(3):489-496. doi: 10.1007/s00246-021-02745-4. Epub 2022 Feb 21. PMID 35190880